CLINICAL TRIAL: NCT02157441
Title: Lower Uterine Compression Sutures for the Treatment of Postpartum Hemorrhage Due to Placenta Previa Complete Centralis; Prospective Study
Brief Title: the Treatment of Postpartum Hemorrhage Due to Placenta Previa Complete Centralis
Acronym: PPH
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, khalid abd aziz mohamed, lecturer of ob/gyn, Benha University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: khalid-ahmed 4
Record Dates: First submitted 2014-06-03; First posted 2014-06-06 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Placenta Previa Complete Centralis
Keywords: Postpartum Hemorrhage; Placenta Previa; uterine cavity
MeSH Terms: conditions — Postpartum Hemorrhage; Placenta Previa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- all patients (Experimental): intervention is lower uterine compression sutures (involved bilateral uterine artery ligation and compression of the lower uterine segment at the same time with one circular stitch) as a conservative treatment for the treatment of postpartum hemorrhage in women with placenta previa complete centralis.
  Interventions: Procedure: lower uterine compression sutures

INTERVENTIONS:
Procedure: lower uterine compression sutures — intervention is lower uterine compression sutures (involved bilateral uterine artery ligation and compression of the lower uterine segment at the same time with one circular stitch) as a conservative treatment for the treatment of postpartum hemorrhage in women with placenta previa complete centralis.

SUMMARY:
Objective: To assess the efficacy of lower uterine compression sutures (involved bilateral uterine artery ligation and compression of the lower uterine segment at the same time with one circular stitch) as a conservative treatment for the treatment of postpartum hemorrhage in women with placenta previa complete centralis. Method: This prospective study of 50 women with postpartum hemorrhage following removal of placenta previa complete centralis during elective cesarean section. All 50 patients will have lower uterine compression sutures (involving bilateral uterine artery ligation and compression of the lower uterine segment at the same time with one circular stitch). All patients will be followed postpartum for evaluation of uterine cavity and menstrual cycles

DETAILED DESCRIPTION:
The investigators conduct a prospective study at Department of Obstetrics and Gynecology, Benha University Hospital, since June 2012 till July 2014, after approval of the study protocol by the Local Ethical Committee.

All patients provide written informed consent to undergo any procedure necessary, including lower uterine compression suturing procedure, as an attempt to avoid hysterectomy. They also provide written informed consent to undergo hysterectomy if all measures attempted to preserve the uterus fail.

All patients have placenta previa (50). The inclusion criteria are a gestation age of ≥ 28 weeks and antepartum hemorrhage; intraoperative postpartum hemorrhage and discovery of a placenta accreta; and an adherent placental part after piecemeal removal of the placenta, with bleeding from the placental site, posterior placenta previa and/or successful piecemeal removal of the placenta.

The first author performed all cesarean deliveries and assisted by the second author. We open the parietal peritoneum by sharp dissection and blunt expansion, high above the bladder, a bladder flap is made and the bladder is retracted. A small median transverse hysterotomy incision is done in the lower uterine segment. It is expanded on both sides using scissors, stopping shortly before the uterine arteries. Active delivery of the placenta is attempted by searching manually for a plane of cleavage between the placenta and the uterus after delivery of the fetus. The study technique comprise lower uterine compression sutures (involved bilateral uterine artery ligation and compression of the lower uterine segment at the same time with one circular stitch).

ELIGIBILITY:
Inclusion Criteria:

* a gestation age of ≥ 28 weeks and antepartum hemorrhage;
* intraoperative postpartum hemorrhage and discovery of a placenta previa;
* successful removal of the placenta

Exclusion Criteria:

* shock due to massive blood loss
* failure of successful removal of the placenta

Ages: 21 Years to 46 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2012-07; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Treatment of Postpartum Hemorrhage | during cesarean section( participants will be followed for the duration of hospital stay)

SECONDARY OUTCOMES:
evaluation of uterine cavity | 6 months after delivery

CONTACTS AND LOCATIONS:
Overall Officials: khalid mohamed, MD, Study Chair — Department of Obstetrics and Gynecology, Benha University Hospital
Locations (1):
- Benha univesity hospital, Banhā, El Qualyobia, Egypt